CLINICAL TRIAL: NCT01540786
Title: An Exploratory Study to Evaluate Bladder Contractions in the Storage Phase (Non Voiding Activities) and Related Bladder Sensation in Healthy Females and Untreated Females With Overactive Bladder ("OAB") Using High Resolution and Conventional Urodynamics
Brief Title: An Exploratory Study to Investigate Bladder Contractions in the Storage Phase and Related Bladder Sensations in Healthy Females and Females With Overactive Bladder (OAB) Using High Resolution and Conventional Urodynamics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It was decided to discontinue the study due to insufficient recruitment
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 905-EC-010
Record Dates: First submitted 2012-02-13; First posted 2012-02-29 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Subjects; Overactive Bladder
Keywords: OAB; High Resolution Urodynamics
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1: OAB subjects (Experimental)
  Interventions: Procedure: High resolution urodynamic assessment; Procedure: Conventional urodynamic assessment
- Part 2: Healthy subjects (Experimental)
  Interventions: Procedure: High resolution urodynamic assessment; Procedure: Conventional urodynamic assessment
- Part 2: OAB subjects (Experimental)
  Interventions: Procedure: High resolution urodynamic assessment; Procedure: Conventional urodynamic assessment

INTERVENTIONS:
Procedure: High resolution urodynamic assessment
Procedure: Conventional urodynamic assessment

SUMMARY:
This study aims to identify differences in bladder contractions during the storage phase (non voiding activities) between OAB subjects and healthy subjects, using high resolution urodynamics.

The study is divided into two parts:

* PART 1: Consists of 5 females with overactive bladder
* PART 2: Consists of 25 females with overactive bladder and 15 healthy females

Part 1 subjects will be enrolled followed by part 2 subjects. The data from part 1 subjects will be reviewed and analysed by a group of experts before starting the second part (part 2) of the study.

DETAILED DESCRIPTION:
The subjects will complete a total of 2 visits and a follow up telephone call (or visit at the investigator's discretion).

Upon meeting eligibility criteria subjects will be screened and complete visit at hospital (Visit 1). They will then be asked to complete procedures such micturition diary, questionnaires and if applicable discontinued their ongoing OAB medication. Upon confirmation of eligibility criteria subjects will then be enrolled and complete visit 2 within 6 to 31 days post V1. At Visit 2 subjects will complete high resolution urodynamic assessment followed by the conventional urodynamic assessment. The visit will take approximately half a day. Safety follow up phone call (or visit at investigator's discretion) will take place 4 to 6 days post visit 2.

ELIGIBILITY:
Inclusion Criteria:

OAB Subjects

* Has history of signs and symptoms of OAB including urinary frequency, urgency or urge incontinence for greater than or equal to 3 months
* At enrolment visit (V2) the subjects must have:

  * At least 1 episode of urgency with or without incontinence in the last 3-day micturition diary
  * Frequency of micturition greater than or equal to 8 per 24 hours period during the 3-day micturition diary period
* At the screening visit, the subject should be either naïve to OAB treatment (e.g no prior history of medications to treat lower urinary tract symptoms (LUTS), including OAB) or currently on treatment for LUTS (including OAB) and is willing to undergo a washout period for 3 weeks

Main Exclusion criteria:

Healthy subjects

* History of lower urinary tract symptoms (LUTS), including OAB
* History of stress urinary incontinence, urethral sphincter incompetence and neurogenic detrusor overactivity
* History of signs or symptoms suggestive of urinary tract infection (confirmed by positive urine analysis)
* History of bladder outlet obstruction (not including detrusor-overactivity) for example bladder/vesicouterine pro-lapse (> grade II) or chronic obstruction
* History of urinary tract surgery less than or equal to 6 months prior to screening
* Has an indwelling catheter or permanent catheter fitted
* History of pelvic area radiotherapy treatment
* Uncontrolled diabetes mellitus
* History of fibromyalgia
* Pregnant or intends to become pregnant during the study or sexually active, of childbearing potential and is unwilling to utilize a reliable method of birth control (note: reliable methods are contraceptive pills of combination type, hormonal implants, injectable contraceptives, sexual abstinence or vasectomized partner)
* Pregnancy within 6 months before screening or breast feeding within 3 months before screening
* History of a positive hepatitis A, B surface antigen, hepatitis C antibody or HIV test result.
* Any use of drugs of abuse within 3 months prior to screening visit.
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to screening visit
* History of drinking more than 14 units of alcohol per week (1 unit = 10 g pure alcohol = 250 ml of beer (5%) or 35 ml of spirits (35%) or 100 ml of wine (12%) within 3 months prior to screening visit
* Is currently receiving or has a history of treatment with alpha blockers, beta receptor blockers or agonists, botulinum toxin (less than 12 months), resiniferatoxin or pelvic floor muscle relaxants less than or equal to 9 months prior to screening

Main exclusion criteria OAB subjects

* Refer to healthy subjects exclusion criteria number 2 to 16

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Identify objective parameters to characterize Non Voiding Activity (NVA) in healthy and OAB subjects using high resolution urodynamic assessment | During the High resolution urodynamics (Day 1)
  NVA is defined as changes of pressure in the bladder lumen. These changes are measured as detrusor pressure (Pdet) calculated from substraction of intra-abdominal pressure (Pabd) from intra-vesical pressure (Pves). All Pdet with an amplitude of at least 1cm of water, frequency below 0.2 Hz and pulse duration between 5 and 60 seconds qualify as NVA.

SECONDARY OUTCOMES:
Identify NVA in healthy and OAB subjects using conventional urodynamic assessment | During High resolution and conventional urodynamic (Day 1) assessments
Assess the subjects bladder sensations measured by visual analogue scale (VAS) and 5-points categorical scale (Appendix 8 & 7) during the high resolution urodynamic and conventional assessments | During High resolution and conventional urodynamic assessments (Day 1)
Assess the correlation between NVA and subjects bladder sensations | During High resolution and conventional urodynamic assessments (Day 1)
Explore NVA in a subgroup of subjects defined by the severity of OAB symptoms collected as background information (3-days bladder diary) | During High resolution and conventional urodynamic assessments (Day 1)
Illustrate the amount of NVA detected with high resolution urodynamic test methodology compared to NVA detected with conventional urodynamic assessments | During High resolution and conventional urodynamic assessments (Day 1)
Assess symptoms severity, bother and its impact on quality of life using: OAB-Q short form and Urogenital Distress Inventory (UDI-6) questionnaires and a 3-Day micturition bladder diary as background information to characterize the study population | During High resolution and conventional urodynamic assessments (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe Ltd.; Principal Investigator, Principal Investigator — Maastricht University Medical Center, Maastricht
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands